CLINICAL TRIAL: NCT04216459
Title: Effect of Anti-inflammatory and Anti-microbial Co-supplementations in Traumatic ICU Patients at High Risk of Sepsis
Acronym: DrNoha-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, lecturer of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: high risk of sepsis
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Major Trauma; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low risk group (No Intervention): no specific treatment will be given
- High risk control (No Intervention): no specific treatment will be given
- High risk DP (Active Comparator): patients will receive one intramuscular (IM) injection of 400,000 IU of cholecalciferol on day- 1 Also, starting from day 1 and till day 6 (for consequential 6 days), patients will receive lactobacillus probiotics (10 billion colony forming unit) in a dose of 6 sachets per day
  Interventions: Drug: oral lactobacillus probiotics plus intramuscular cholecalciferol
- High risk CB (Active Comparator): Patients will receive vitamin C plus thiamine starting from day 1 in a dose of 1 gm vitamin C and 200 mg thiamine intravenous 4 times at 12-hour intervals for 48 hours
  Interventions: Drug: intravenous vitamin C plus thiamine

INTERVENTIONS:
Drug: oral lactobacillus probiotics plus intramuscular cholecalciferol — According to leukocyte anti- sedimentation rate (LAR) result on day 1 patients will be classified into high risk for sepsis patients (LAR < 15 %) and low risk for sepsis patients (LAR ≥ 15%) High risk sepsis patients will be randomly allocated into one of the 3 groups (sealed opaque envelops) to vitamin D plus probiotics intervention group (HR-DP) group. to vitamin C plus vitamin B intervention group (HR-CB) group. to control group (HR-C) group that does not receive any supplement
  Arms: High risk DP
Drug: intravenous vitamin C plus thiamine — starting from day 1 in a dose of 1 gm vitamin C and 200 mg thiamine intravenous 4 times at 12-hour intervals for 48 hours
  Arms: High risk CB

SUMMARY:
The occurrence of sepsis in trauma patients is a very serious complication. Identifying trauma patients at high risk of sepsis was not revealed in the latest surviving sepsis campaign in 2016. Several biomarkers have been proposed for early prediction of sepsis in trauma patients as leukocyte anti sedimentation rate (LAR) and the proinflammatory cytokine monocyte chemo attractant protein-1 (MCP-1). Sepsis prophylaxis before occurrence of multi-organ failure still represents a major challenge. Vitamin D and probiotics have antimicrobial, anti-inflammatory and gut microbiota immune modulatory properties.Little is known about the effect of vitamin D and probiotics co-supplementation on the inflammatory response in trauma patients at high risk of sepsis.

Another promising strategy is the use of vitamin C in addition to thiamine. Trauma is associated with increased oxidative stress and vitamin C deficiency. High dose vitamin C is required to restore oxidant-antioxidant balance. Vitamin C and thiamine have shown promising results in treatment of sepsis. Vitamin C possesses anti-inflammatory, endothelial protective and anti-microbial effects. Thiamine is the precursor of thiamine pyrophosphate (TPP), a key enzyme in Krebs cycle.

DETAILED DESCRIPTION:
This study will investigate effect of vitamin D and probiotics versus Vitamin C and thiamine on inflammatory response (represented by change in MCP-1 level), Sequential Organ Failure Assessment (SOFA) Score and Acute Physiology and Chronic Health Evaluation II (APACHE II) in trauma patients at high risk of sepsis. Secondary goal is to assess if the predictive ability of MCP-1 plus LAR to determine high risk of sepsis in major trauma intensive care patients and if there is correlation between LAR and MCP-1.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients admitted to ICU within 24 hours from trauma onset with injury severity score (ISS) ≥ 16 will be recruited after obtaining informed consent

Exclusion Criteria:

* • Patients admitted to ICU after time exceeding 24 hours from trauma onset.

  * Patients whose age is less than 18 years.
  * Pregnant female.
  * Breast feeding women.
  * Arrest within 24 hours of admission.
  * Immune deficiency or administration of immune suppressant drugs.
  * Serum calcium greater than or equal to 10 mg/dl or phosphate greater than or equal 6 mg/dl.
  * History of primary parathyroid disease.
  * Metabolic bone disease.
  * Sarcoidosis.
  * End stage renal disease.
  * receiving intermittent renal replacement therapy (RRT).
  * Failure of enteral feeding or any contraindication to enteral administration.
  * Obesity , body mass index (BMI > 35 kg/m2)
  * Known contraindication to vitamin C or thiamine (oxalate nephropathy or known glucose-6-phosphate dehydrogenase deficiency)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | 0n the Day 0-Day 6 from onset of trauma
  minim 0 maximum 71 Increasing score is associated with increasing risk of ICU mortality

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | 0n the Day 0-Day 6 from onset of trauma
  minim 0 maximum 24 The acute increase of 2 or more in SOFA points indicates sepsis
Monocyte chemo attractant protein 1 (MCP-1) | 0n the Day 0-Day 6 from onset of trauma
  Optimum cut-off value of MCP-1 for prediction of sepsis in severe trauma ICU patients is 240.7 pg/ml The decrease in its level indicates less inflammatory response and better patient out comes

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ahmed Abozeid, MD, Study Director — Faculty of Medicine - Mansoura University
Locations (1):
- Mansoura University-Emergency hospital-ICU, Al Mansurah, Egypt

REFERENCES:
- [Derived] Kamel NA, Soliman MM, Abo-Zeid MA, Shaaban MI. Effect of Anti-Inflammatory and Antimicrobial Cosupplementations on Sepsis Prevention in Critically Ill Trauma Patients at High Risk for Sepsis. Front Pharmacol. 2021 Nov 29;12:792741. doi: 10.3389/fphar.2021.792741. eCollection 2021. PMID 34912231